CLINICAL TRIAL: NCT05612568
Title: Five Years of Eye Screening for Amblyopia Risk Factors in Children Aged <3 Years in Flanders: Epidemiological Retrospective Study
Brief Title: 5 Years of Eye Screening for ARF in Children Aged <3 Years in Flanders
Status: Active, not recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S64110
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Researchers will investigate the distribution and evolution of amblyopia risk factors and other refractive errors in children younger than 3 years of age. The significance and magnitude of current global evolutions in ARF and refractive errors will be verified to update current guidelines and practices. Better insight in associated factors of amblyopia risk factors will contribute to current understanding of amblyopia.

DETAILED DESCRIPTION:
The eye screening program of the Flemish governmental agency 'Kind en Gezin' is a well-implemented screening program for detection of ARF in children under the age of 3 years. This screening covers almost 85% of all children born in the Flemish community. Valuable information about distribution and determinants of refractive errors and ARF are collected at 'Kind en Gezin', but remain unstudied until today.

The aim is to analyze the distribution and evolution of refractive errors in children under the age of 3 years in Flanders. One supposes that identification of patterns in this distribution, and identification of determinants that influence ARF, will lead to improved knowledge about amblyopia (risk factors) and on their turn help optimize the ARF screening program. Evaluation of the distribution and evolution of refractive errors over time, and comparison with global results, will also give researchers insight in the significance of the myopia epidemic in Flanders.

ELIGIBILITY:
Inclusion Criteria:

* We include all children with a PlusOptix screening between 2013 and 2018 with the age of 12±1 months or 30±1 months. Children who were screened twice, can be included twice with both screening results.

Exclusion Criteria:

* none

Ages: 13 Months to 31 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We include all children with a PlusOptix screening between 2013 and 2018 with the age of 12±1 months or 30±1 months.
Sampling Method: Probability Sample
Enrollment: 250000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Refractive error per eye | Day 1
  Sphere, cylinder, spherical equivalent
Difference in refractive error between both eyes | Day 1
  Sphere OD-OS, cylinder OD-OS, spherical equivalent OD-OS

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No